CLINICAL TRIAL: NCT03753438
Title: Intragastric Balloon in Compensated NASH(Non Alcoholic Steato Hepatitis) Cirrhotics-An Observational Study
Brief Title: Intragastric Balloon in Compensated NASH(Non Alcoholic Steato Hepatitis) Cirrhotics
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-NASH-04
Record Dates: First submitted 2018-10-17; First posted 2018-11-27 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intragastric Balloon: Intragastric Balloon will be placed for 6 months
  Interventions: Procedure: Intragstric Ballooning

INTERVENTIONS:
Procedure: Intragstric Ballooning — Intragstric Ballooning will be put.

SUMMARY:
The study will be conducted in department of Hepatology at ILBS, the patients will be recruited from the OPD or IPD . The obese cirrhotic patients with NASH will be observed for standard of care and also patients who undergo IGB placement as part of weight reduction policy in these group of patients and will undergo an UGI endoscopy followed by placement of intragastric balloon. Then the patients will be admitted for 2-3 days and followed up till 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18 and 65 years
* NASH (Non Alcoholic SteatoHepatitis) cirrhosis
* BMI > 30 and failure to control weight despite full dietary and life style modifications.
* Compensated : CTP 6 & 7 without any evidence of decompensation in form of Hepatic encephalopathy, ascites, GI bleed or prolonged jaundice.
* Small varices: Grade I varices

Exclusion Criteria:

* Alcoholic liver disease
* Advanced liver disease with ascites, hepatic encephalopathy
* Other liver diseases such as chronic hepatitis B, chronic hepatitis C, Wilsons' disease, Hemochromatosis, glycogen storage diseases etc.
* Pregnancy
* Unwilling patients
* Large varices
* Past h/o GI bleed
* Hiatus hernia
* Gastric ulcer
* Severe esophagitis (Grade B and above)
* Severe PHG or gastric erythema

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NASH (Non Alcoholic SteatoHepatitis) cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change in weight from baseline | 3 months
Change in weight reduction from baseline | 6 Months

SECONDARY OUTCOMES:
Change in development of liver related complications | 3 Months
Change in development of liver related complications | 6 Months
Improvement of insulin resistance in both groups. | 3 Months
Improvement of insulin resistance in both groups. | 6 Months
Decreased usage of medications for diabetes mellitus in both groups. | 3 Months
Decreased usage of medications for diabetes mellitus in both groups. | 6 Months
Decreased usage of medications for HOMA-IR (Homeostatic Model Assessment-Insulin Resistance) in both groups. | 3 Months
Decreased usage of medications for HOMA-IR (Homeostatic Model Assessment-Insulin Resistance) in both groups. | 6 Months
Improvement of insulin resistance and decreased usage of medications for TNF-α (Tumor Necrosis Factor-Alpha). | 3 Months
Improvement of insulin resistance and decreased usage of medications for TNF-α (Tumor Necrosis Factor-Alpha). | 6 Months
Improvement in liver parameters such as serum albumin in both groups. | 3 Months
Improvement in liver parameters such as serum albumin in both groups. | 6 Months
Improvement liver parameters such as INR in both groups | 3 Months
Improvement in liver parameters such as INR in both groups. | 6 Months
Improvement in liver parameters such as bilirubin in both groups | 3 Months
Improvement in liver parameters such as bilirubin in both groups. | 6 Months
Disappearance of esophageal varices in both groups. | 3 Months
Disappearance of esophageal varices in both groups. | 6 Months
Improvement in LSM (liver stiffness on fibroscan) in both groups | 3 Months
Improvement in LSM (liver stiffness on fibroscan) in both groups. | 6 Months
Improvement in CAP (Controlled Attenuation Index) in both groups. | 3 Months
Improvement in CAP (Controlled Attenuation Index) in both groups. | 6 Months
Improvement in HVPG (Hepatic venous Pressure Gradient) in both groups. | 3 Months
Improvement in HVPG (Hepatic venous Pressure Gradient) in both groups. | 6 Months
Improvement in liver histology post completion of study in both groups. | 6 Months
Change in hormonal levels such as Adiponectin level in both groups.. | 3 Months
Change in hormonal levels such as Adiponectin level in both groups. | 6 months
Change in hormonal levels such as leptin level in both groups. | 3 Months
Change in hormonal levels such as Ghrelin level in both groups.. | 3 Months
Change in hormonal levels such as Ghrelin level in both groups.. | 6 Months
Change in hormonal levels such as Endothelin level in both groups.. | 3 Month
Change in hormonal levels such as Endothelin level in both groups.. | 6 Month

CONTACTS AND LOCATIONS:
Overall Officials: Shiv Kumar Sarin, DM, Principal Investigator — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vijayaraghavan R, Sarin SK, Bharadwaj A, Anand L, Maiwall R, Choudhury A, Benjamin J, Kanal U, Jamwal KD. Intragastric Balloon in Obese Compensated Nonalcoholic Steatohepatitis Cirrhosis Patients Is Safe and Achieves Significant Weight Reduction at 6-Months. Dig Dis Sci. 2023 Mar;68(3):1035-1041. doi: 10.1007/s10620-022-07596-4. Epub 2022 Jun 28. PMID 35763235